CLINICAL TRIAL: NCT00529854
Title: Surgical and Trauma Intensive Care Unit Documentation and Billing Improvements With Medical Informatics
Brief Title: SIC-IR Billing and Documentation
Acronym: SIC-IR
Status: Completed | Type: Observational
Sponsor: MetroHealth Medical Center (Other)
Other Study IDs: IRB07-00922
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2008-02-27 (Estimated); Status verified 2008-02

CONDITIONS: Medical Record Documenation; Surgical and Trauma Intensive Care Unit Billing
Keywords: Intensive care unit; medical documentation; medical billing

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Observational evaluation of current billing and documentation practices
- 2: Use of SIC-IR Billing Module
  Interventions: Other: SIC-IR Billing Module

INTERVENTIONS:
Other: SIC-IR Billing Module — Medical informatic application designed to help with billing and documentation within the surgical and trauma intensive care unit
  Groups: 2

SUMMARY:
Accurate documentation in the patient medical record is critical to ensure proper diagnosis coding and subsequent hospital reimbursement. Multiple studies have demonstrated that clinicians often omit diagnoses which may result in insurance company denials and significant delays in payment. In addition, omitting diagnoses decreases the severity of patient illness which is often used as a risk adjustment tool to compare institution and physician outcomes. Medical informatics has been used to help improve accurate diagnosis documentation as well as improve billing efficiency. We plan to utilize a medical informatics program called SIC-IR (Surgical Intensive Care - Infection Registry) to improve documentation and attending billing efficiency within the surgical and trauma intensive care unit (STICU). We propose a six month study: a three month observational evaluation of current billing procedures followed by a three month prospective evaluation using a newly created SIC-IR billing module. The outcome measures will include the number of ICD-9 and CPT codes at discharge per patient, severity of patient illness based on documentation, STICU charges, number of insurance company denials, DRG relative weights, as well as a qualitative assessment of attending physician use of the electronic billing module. The observational and prospective patient populations will be compared for total patient-days in the STICU, ventilator-days, antibiotic-days, infectious complications per patient, and injury severity score (trauma patients only) to ensure the populations are similar and only the documentation and billing changes can account for our measured outcomes. We hypothesize that the SIC-IR billing module will increase the number of patient ICD-9 and CPT codes at discharge, increase severity of STICU patient illness via accurate documentation, increase total STICU charges, decrease insurance company denials, and be an efficient and well accepted electronic medical application.

DETAILED DESCRIPTION:
1. An observational evaluation will be performed for all STICU patients over a three month time period.

   1. Data collected will be the outcome measures listed above (Number of ICD-9 codes at discharge, number of CPT codes at discharge, ext)
   2. In addition the total number of STICU patient-days, ventilator-days, central line-days, confirmed infectious complications, injury severity scores for trauma patients, and antibiotic-days will be collected over the three month period. This will serve as a way to ensure the observational and prospective populations are not different, and only the documentation and billing methods changed.
2. The SIC-IR billing module will be released on October 1st, 2007 after attending physician training on its use.
3. A prospective evaluation will be performed for all STICU patients over a three month time period

   1. Data collected will be the outcome measures listed above (Number of ICD-9 codes at discharge, number of CPT codes at discharge, ext)
   2. In addition the total number of STICU patient-days, ventilator-days, central line-days, confirmed infectious complications, injury severity scores for trauma patients, and antibiotic-days will be collected over the three month period. This will serve as a way to ensure the observational and prospective populations are not different, and only the documentation and billing methods changed.
4. After the 3 month prospective evaluation, the attending physicians will be given a survey to document their acceptance or rejection of the billing module.
5. The observational and prospective documentation and billing data will be compared.

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients admitted to the surgical and trauma intensive care unit a a single level one trauma center care for by the surgical intensivist

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All surgical and trauma intensive care unit patients addmitted to our reional Level I trauma center
Enrollment: 814 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Number of ICD-9 codes at discharge (per patient) | 6 months
Number of STICU specific ICD-9 codes at discharge (per patient) | 6 months
Number of CPT codes at discharge (per patient) | 6 months
Number of STICU specific CPT codes at discharge (per patient) | 6 months
Number of specific evaluation and management codes used (per patient) | 6 months
Total STICU charges at discharge (per patient) | 6 months
Number of denied insurance claims (per month) | 6 months
Estimated patient survival based on documentation (illness severity) (per patient) | 6 months
DGR relative weight at discharge (per patient) | 6 months
Qualitative assessment of attending approval of the SIC-IR module | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Golob, MD, Study Director — MetroHealth Medical Center; Jeffrey A Claridge, MD, Principal Investigator — MetroHealth Medical Center; Adam MA Fadlalla, PhD, Study Director — Cleveland State University
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States